CLINICAL TRIAL: NCT06539065
Title: The Effects of VR Interactive Games on Balance and Quality of Life Enhancement for Elderly in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: N202210004
Record Dates: First submitted 2023-06-29; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2023-06

CONDITIONS: Virtual Reality
Keywords: VR; Balance; Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): The experimental group received a twelve-week intervention of 36 sessions using VR interactive games in their exercise prescription
  Interventions: Device: VR interactive games
- Non-VR group (No Intervention): control group followed the original instructor-led exercise intervention as the course content.

INTERVENTIONS:
Device: VR interactive games — The experimental group received a twelve-week intervention of 36 sessions using VR interactive games in their exercise prescription,
  Arms: VR group

SUMMARY:
The goal of this clinical trial is to learn about the effectiveness of the incorporating VR interactive games into exercise courses of the elderly in the community.The main questions It aims to answer are: can It improve their balance ability and the quality of life.

Participants will receive a Twelve-week intervention of 36 sessions using VR interactive games in their exercise prescription, While the control group will follow the original iInstructor-led exercise intervention as the course content.

DETAILED DESCRIPTION:
Both groups will undergo three sessions per week, one hour per session, for a total of 12 weeks and 36 sessions of intervention. Before and after competing all sessions, the effectiveness of this intervention will be assessed.

Some physical assessments will be done by all participants such as 2-minute step, right chair sit and reach, left chair sit and reach to compare if any difference between two groups. and participants will do a questionaire to evaluate the psychological and environmental quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 or above
2. Capable of communicating in Mandarin or Taiwanese, and willing to participate in interviews or complete questionnaires
3. Free of mobility impairments

Exclusion Criteria:

1. Stroke with sequelae of mobility impairments
2. Parkinson's disease
3. Motor neurone disease
4. Severe Cardio-vascular disease
5. Degenerative joint disease with flare-ups in past three months
6. With a lower limb joint surgery in past 3 months
7. Vertigo

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Balance ability | Physical assessment done 2 weeks before and 2 weeks after 12 weeks courses
  The scores of five physical assessments
Life quality | Questionnaire done 2 weeks before and 2 weeks after 12 weeks courses
  The score of questionnaire done by all participants

CONTACTS AND LOCATIONS:
Overall Officials: Chueh-Ho Lin, PhD, Study Chair — Taipei Medical University
Locations (1):
- Taipei medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
the datasets generated in this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the datasets generated in this study are available from the corresponding author upon reasonable request.
Access Criteria: no criteria

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT06539065/Prot_SAP_ICF_000.pdf